CLINICAL TRIAL: NCT07264348
Title: Effects of a 4-month Intervention on Cardiometabolic, Hormonal, Inflammatory, Liver, Renal, Electrolyte, and Muscle Enzyme Parameters in Pre- and Post-Menopausal Overweight and Obese Women: A Randomized Controlled Trial
Brief Title: Cardiometabolic and Hormonal Adaptations to 4-Month Zumba Training in Overweight/Obese Women
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: High Institute of Sports and Physical Education of Kef (Other)
Responsible Party: Principal Investigator, Wissal Abassi, Principal Investigator, High Institute of Sports and Physical Education of Kef
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HORMONE-2025
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Hormone; Cardiovascular; Obesity & Overweight
Keywords: Overweight; Obesity; Pre-menopause; Post-menopause; Zumba Training; Cardiometabolic Health; Hormonal Adaptations; Lipid Profile
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental Group 1:Pre-menopausal (Experimental): performed Zumba training, 4 × 60 min/week, 4 months
  Interventions: Behavioral: Zumba training
- Control Group 1 (No Intervention): No training intervention was intended for the control group.
- Experimental Group 2:Post-menopausal (Experimental): performed Zumba training, 4 × 60 min/week, 4 months
  Interventions: Behavioral: Zumba training
- Control group 2 (No Intervention): No training intervention was intended for the control group.

INTERVENTIONS:
Behavioral: Zumba training — Participants assigned to the experimental groups will perform a supervised Zumba training program for 10 weeks, with 4 sessions per week, each session lasting 60 minutes. Sessions will include a standardized warm-up (10 minutes), choreographed dance-based aerobic sequences performed at moderate intensity (40 minutes), and a cool-down with stretching (10 minutes).
  Arms: Experimental Group 1:Pre-menopausal; Experimental Group 2:Post-menopausal

SUMMARY:
This study aims to evaluate the effects of a 4 month Zumba training program on cardiometabolic, hormonal, inflammatory, hepatic, renal, and functional parameters in overweight and obese women. Participants will be classified according to menopausal status (pre- or post-menopausal) and randomly assigned to an exercise group or a non-exercise control group.

DETAILED DESCRIPTION:
Overweight and obesity are associated with metabolic dysregulation, hormonal imbalance, chronic inflammation, and reduced physical capacity. Zumba training is a dance-based aerobic exercise that can improve cardiovascular fitness, energy expenditure, and adherence to physical activity programs.

This study will assess the effects of a 4 month Zumba training program (4 sessions per week, 60 minutes per session) on: Body composition and anthropometric measures, Aerobic capacity, Hormonal profile, Lipid profile, Inflammatory biomarkers, Liver enzymes, Renal function markers, Electrolytes, Muscle enzymes, Pre- and post-training measurements will be taken under standardized conditions.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18-65 years
* BMI ≥ 25 kg/m²
* Pre-menopausal or post-menopausal (classified clinically)
* Voluntary written informed consent

Exclusion Criteria:

* Hormonal therapy or weight-loss medications
* Endocrine diseases or chronic illness
* Recent intense physical training (<48 hours before baseline)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 73 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Body Mass Index (BMI) | Baseline and after 4 months of Zumba intervention.
  BMI calculated as weight (kg) divided by height squared (m²).
Body Fat Percentage | Baseline and after 4 months of Zumba intervention.
  Total body fat measured by digital scale (Tanita BC-533).
Waist Circumference | Baseline and after 4 months of Zumba intervention.
  Measured at the narrowest point between the rib cage and iliac crest using a tape measure.
Waist-Hip Ratio | Baseline and after 4 months of Zumba intervention.
  Calculated by dividing waist circumference by hip circumference.
Hip Circumference | Baseline and after 4 months of Zumba intervention.
  Measured at the widest point of the hips using a tape measure.
Prolactin | Baseline and after 4 months of the intervention.
  Serum prolactin concentration (ng/mL).
Testosterone | Baseline and after 4 months of the intervention.
  Serum testosterone concentration (ng/dL).
Cortisol | Baseline and after 4 months of the intervention.
  Serum cortisol concentration (µg/dL).
Progesterone | Baseline and after 4 months of the intervention.
  Serum progesterone concentration (ng/mL).
Estradiol | Baseline and after 4 months of the intervention.
  Serum estradiol concentration (pg/mL).
Follicle-Stimulating Hormone (FSH) | Baseline and after 4 months of the intervention.
  Serum FSH concentration (mIU/mL).
Luteinizing Hormone (LH) | Baseline and after 4 months of the intervention.
  Serum LH concentration (mIU/mL).
Thyroid Stimulating Hormone (TSH) | Baseline and after 4 months of the intervention.
  Serum TSH concentration (µIU/mL).
Free Thyroxine (FT4) | Baseline and after 4 months of the intervention.
  Serum free T4 concentration (ng/dL).
Parathyroid Hormone (PTH) | Baseline and after 4 months of the intervention.
  Serum PTH concentration (pg/mL).
Total Cholesterol | Baseline and after 4 months of the intervention.
  Serum total cholesterol concentration (mg/dL).
High-Density Lipoprotein (HDL) Cholesterol | Baseline and after 4 months of the intervention.
  Serum HDL cholesterol concentration (mg/dL).
Low-Density Lipoprotein (LDL) Cholesterol | Baseline and after 4 months of the intervention.
  Serum LDL cholesterol concentration (mg/dL).
Triglycerides | Baseline and after 4 months of the intervention.
  Serum triglyceride concentration (mg/dL).
C-Reactive Protein (CRP) | Baseline and after 4 months of the intervention.
  Serum CRP concentration (mg/L).
Erythrocyte Sedimentation Rate (ESR) | Baseline and after 4 months of the intervention.
  ESR measured in mm/hr.
Complete Blood Count (CBC) | Baseline and after 4 months of the intervention.
  Includes neutrophils, lymphocytes, monocytes, eosinophils, basophils (cells/µL).
Alanine Aminotransferase (ALT) | Baseline and after 4 months of the intervention.
  Serum ALT concentration measured in U/L.
Aspartate Aminotransferase (AST) | Baseline and after 4 months of the intervention.
  Serum AST concentration measured in U/L.
Alkaline Phosphatase (ALP) | Baseline and after 4 months of the intervention.
  Serum ALP concentration measured in U/L.
Gamma-Glutamyl Transferase (GGT) | Baseline and after 4 months of the intervention.
  Serum GGT concentration measured in U/L.
Lactate Dehydrogenase (LDH) | Baseline and after the 4 months of the intervention.
  Serum LDH concentration measured in U/L.
Gamma-Glutamyl Transferase (GGT) | Baseline and after the 4 months of the intervention.
  Serum GGT concentration measured in U/L.
Bilirubin Total | Baseline and after the 4 months of the intervention.
  Total serum bilirubin concentration measured in mg/dL.
Bilirubin Direct | Baseline and after the 4 months of the intervention.
  Direct (conjugated) serum bilirubin concentration measured in mg/dL.
Creatinine | Baseline and after 4 months of the intervention.
  Serum creatinine concentration measured in mg/dL, indicator of kidney function.
Urea | Baseline and after 4 months of the intervention.
  Serum urea concentration measured in mg/dL, indicator of kidney function.
Uric Acid | Baseline and after 4 months of the intervention.
  Serum uric acid concentration measured in mg/dL, indicator of kidney function.
Sodium (Na) | Baseline and after 4 months of the intervention.
  Serum sodium concentration measured in mmol/L.
Potassium (K) | Baseline and after 4 months of the intervention.
  Serum potassium concentration measured in mmol/L.
Calcium (Ca) | Baseline and after 4 months of training.
  Serum calcium concentration measured in mg/dL.
Magnesium (Mg) | Baseline and after 4 months of training.
  Serum magnesium concentration measured in mg/dL.
Phosphate (PO₄) | Baseline and after 4 months of training.
  Serum phosphate concentration measured in mg/dL.
Creatine Phosphokinase (CPK) | Baseline and after 4 months of training.
  Serum CPK concentration measured in U/L, indicator of muscle damage.
Lactate Dehydrogenase (LDH) | Baseline and after 4 months of training.
  Serum LDH concentration measured in U/L, indicator of muscle and tissue damage.

SECONDARY OUTCOMES:
Resting Heart Rate | Baseline and after 4 months of Zumba intervention.
  Measured using automated device (Omron BP652).
Blood Pressure (Systolic and Diastolic) | Baseline and after 4 months of Zumba intervention.
  Measured using an automated arm cuff (Omron BP652).
6-Minute Walk Test (6MWT) Distance | Baseline and after 4 months of Zumba intervention.
  Distance walked in 6 minutes on a 30-meter straight corridor.

CONTACTS AND LOCATIONS:
Overall Officials: Wissal abassi, Principal Investigator — Research Unit "Sport Sciences, Health and Movement"(UR22JS01) High Institute of Sport and Physical Education of Kef, University of Jendouba, 7100 Kef, Tunisia.

IPD SHARING:
Plan to Share IPD: No
For confidentiality reasons, all data from this study will be available upon request.